CLINICAL TRIAL: NCT02564211
Title: A Phase III, Multicenter, Open-label Long-term Treatment Trial to Assess the Safety and Efficacy of Addition of Ipragliflozin in Japanese Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Sitagliptin Monotherapy in Addition to Diet and Exercise Therapy
Brief Title: Ipragliflozin Add-on Long-term Study in Japanese Participants With Type 2 Diabetes Mellitus on Sitagliptin (MK-0431J-849)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0431J-849; 153083 (Registry Identifier: JAPIC-CTI); MK-0431J-849 (Other: Merck)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Results first posted 2018-03-14 (Actual); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — ipragliflozin; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ipragliflozin (Experimental): Ipragliflozin one 50 mg tablet co-administered with one 50 mg sitagliptin once daily (QD) for 52 weeks in addition to diet and exercise therapy.
  Interventions: Drug: Ipragliflozin; Drug: Sitagliptin

INTERVENTIONS:
Drug: Ipragliflozin — one 50 mg tablet QD
Drug: Sitagliptin — one 50 mg tablet QD

SUMMARY:
This is a study to assess the safety and efficacy of the addition of ipragliflozin to sitagliptin in Japanese participants with Type 2 diabetes mellitus (T2DM) who have inadequate glycemic control on sitagliptin, diet, and exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

* Has Type 2 diabetes mellitus
* Has inadequate glycemic control on diet/exercise therapy and sitagliptin monotherapy
* Hemoglobin A1C (HbA1c) ≥7.0% and ≤10.0% before study participation

Exclusion Criteria:

* History of type 1 diabetes mellitus or a history of ketoacidosis
* History of any of the following medications: Thiazolidinediones (TZD) and/or insulin within 12 weeks prior to study participation, sodium glucose cotransporter 2 (SGLT2) inhibitors anytime
* Currently has a urinary tract infection or genital infection with subjective symptom

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2015-10-26 (Actual); Primary Completion 2017-03-07 (Actual); Study Completion 2017-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Kaku K, Kadowaki T, Seino Y, Okamoto T, Shirakawa M, Sato A, O'Neill EA, Engel SS, Kaufman KD. Efficacy and safety of ipragliflozin in Japanese patients with type 2 diabetes and inadequate glycaemic control on sitagliptin. Diabetes Obes Metab. 2021 Sep;23(9):2099-2108. doi: 10.1111/dom.14448. Epub 2021 Jun 15. PMID 34033212

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ipragliflozin
Started | 77
Completed | 73
Not Completed | 4
Not completed — Adverse Event | 4

BASELINE CHARACTERISTICS:
Arm/Group | Ipragliflozin
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 77
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
HbA1c [Mean (Standard Deviation); unit: Percentage] | 8.01 (0.69)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experienced at Least 1 Adverse Event (AE)
Description: An AE was any unfavorable or unintended sign, symptom, or disease, and a causal relationship to the relevant investigational product is not considered. An AE could therefore be any unfavorable and unintended sign, including results from laboratory assessments, physical examination, electrocardiograms, and vital sign assessments. The percentage of participants that had AE was recorded.
Time Frame: Up to 54 weeks
Population: All participants who received at least 1 dose of treatment period study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Ipragliflozin
Number analyzed (Participants) | 77
Percentage of participants | 77.9

2. Primary Outcome: Percentage of Participants Who Had Study Drug Discontinued Due to an AE
Description: The percentage of participants who had study treatment stopped due to an AE regardless if they completed study.
Time Frame: Up to 52 weeks
Population: All participants who received at least 1 dose of treatment period study medication.
Measure: Number; unit: Percentage of Participants
Arm/Group | Ipragliflozin
Number analyzed (Participants) | 77
Percentage of Participants | 5.2

3. Secondary Outcome: Change From Baseline in HbA1c
Description: Participants had HbA1c levels determined at baseline and at Week 52. HbA1c is reported as a percentage. A negative number reflects a decrease in percentage.
Time Frame: Baseline and Week 52
Population: All participants who received at least 1 dose of treatment period study medication. had at least 1 measurement of the outcome variable (baseline or post-baseline) and had baseline data for those analyses that required baseline data.
Measure: Mean (95% Confidence Interval); unit: Percent
Arm/Group | Ipragliflozin
Number analyzed (Participants) | 73
Percent | -0.80 [-0.96 to -0.65]

ADVERSE EVENTS:
Time Frame: Up to 54 weeks
Description: All participants that received at least 1 dose of study drug.
Groups:
- Ipragliflozin 50 mg: Ipragliflozin one 50 mg tablet co-administered with one 50 mg sitagliptin once daily (QD) for 52 weeks in addition to diet and exercise therapy.
Arm/Group | Ipragliflozin 50 mg
All-Cause Mortality (participants affected / at risk) | 0/77
Serious Adverse Events (participants affected / at risk) | 5/77
Other Adverse Events (participants affected / at risk) | 44/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipragliflozin 50 mg (N=77)
Angina pectoris (Cardiac disorders) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ipragliflozin 50 mg (N=77)
Constipation (Gastrointestinal disorders) | 6 (6)
Thirst (General disorders) | 8 (8)
Influenza (Infections and infestations) | 5 (5)
Nasopharyngitis (Infections and infestations) | 22 (33)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12)
Pollakiuria (Renal and urinary disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-05): https://cdn.clinicaltrials.gov/large-docs/11/NCT02564211/Prot_SAP_000.pdf